CLINICAL TRIAL: NCT00303888
Title: A Randomized Placebo-Controlled Phase Ib/IIa Safety, Tolerability and Efficacy Study of Oral Phenoxodiol in Combination With Docetaxel Versus Docetaxel Alone in Patients With Recurrent Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Brief Title: Docetaxel With or Without Phenoxodiol in Treating Patients With Recurrent Advanced Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cavity Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0504027640; YALE-HIC-27640; YALE-012705
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; recurrent primary peritoneal cavity cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; stage IV primary peritoneal cavity cancer; recurrent fallopian tube cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Docetaxel; phenoxodiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive docetaxel IV over 1 hour on days 1, 8, and 15 and oral placebo three times daily on days 1-21.
  Interventions: Drug: docetaxel; Other: placebo
- Arm II (Experimental): Patients receive oral phenoxodiol three times daily on days 1-21 and docetaxel IV over 1 hour on days 1, 8, and 15.
  Interventions: Drug: docetaxel; Drug: idronoxil

INTERVENTIONS:
Drug: docetaxel — Given IV
Drug: idronoxil — Given orally
  Arms: Arm II
Other: placebo — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Phenoxodiol may help docetaxel work better by making tumor cells more sensitive to the drug.

PURPOSE: This randomized phase I/II trial is studying the side effects of docetaxel when given together with either phenoxodiol or placebo and to see how well it works in treating patients with recurrent advanced ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of combination therapy comprising phenoxodiol and docetaxel in patients with recurrent or persistent advanced ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer.

Secondary

* Determine the effect of phenoxodiol on the toxicity of docetaxel using a weekly treatment regimen.
* Determine if combination therapy comprising phenoxodiol and docetaxel is more efficacious than docetaxel therapy alone.
* Determine if combination therapy comprising phenoxodiol and docetaxel affects blood levels of either drug.
* Determine phenotypic differences in the tumor cells of "responders" and "non-responders."

OUTLINE: This is a randomized, placebo-controlled, double-blind study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on days 1, 8, and 15 and oral placebo three times daily on days 1-21.
* Arm II: Patients receive oral phenoxodiol three times daily on days 1-21 and docetaxel as in arm I.

Treatment in both arms repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed monthly for 6 months, every 3 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

3/31/2017 NOTE

This study was terminated 10/2009 due to lack of enrollment. The study never progressed to Phase 2.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Ovarian epithelial cancer
  * Fallopian tube cancer
  * Primary peritoneal cavity cancer
* Recurrent advanced disease

  * Eligible for second-line to fifth-line chemotherapy
  * Received platinum and taxane combination chemotherapy as first-line treatment with disease recurrence > 6 months after conclusion of therapy

    * No demonstrated refractoriness or resistance to weekly docetaxel
* Meets 1 of the following criteria:

  * Doubling of blood levels of CA125 in the past 6 months and CA125 levels ≥ 2 times upper limit of normal (ULN)
  * Measurable disease defined as ≥ 1 lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* No active CNS metastases

  * Prior CNS metastases allowed provided they were treated with radiation therapy and disease has been stable for 4 weeks

PATIENT CHARACTERISTICS:

* Karnofsky performance score ≥ 60%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Life expectancy ≥ 3 months
* Creatinine ≤ 1.5 mg/dL
* Transaminases ≤ 3 times upper limit of normal (ULN)
* Bilirubin normal
* Platelet count > 100,000/mm^3
* WBC > 3,000/mm^3
* Neutrophil count > 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Peripheral neuropathy ≤ grade 1
* Relative proportions of AST, ALT, and alkaline phosphatase according 1 to the following criteria:

  * Alkaline phosphatase (AP) normal AND AST/ALT ≤ 5 times ULN
  * AP ≤ 2.5 times ULN AND AST/ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST/ALT normal
* No active infection
* No concurrent severe and/or uncontrolled medical disease (e.g., uncontrolled diabetes, hypertension, ischemic heart disease, or congestive heart failure)
* No history of chronic active hepatitis or cirrhosis
* No history of severe hypersensitivity to docetaxel or other drugs formulated with polysorbate 80

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No investigational agents within 4 weeks prior to study entry
* Recovered from prior antineoplastic therapy
* No other concurrent investigational drugs
* No other concurrent chemotherapy, radiotherapy, immunotherapy, or hormonal antitumor therapy

  * Concurrent localized radiation therapy allowed for control of local disease complications (e.g., bone metastases) that do not represent a general progression of the disease status
* No concurrent grapefruit or grapefruit juice
* No concurrent amifostine

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Survival (progression-free/recurrence-free interval and overall survival)
Tumor response as assessed by RECIST criteria and clinical examination
Changes in tumor marker CA125 as assessed by Rustin criteria
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Rutherford, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No